CLINICAL TRIAL: NCT00235989
Title: An Open-label Extension Study of the Double-blind, Randomized, Parallel Group, Multicenter Phase 2 Study 307000A to Further Evaluate the Safety and Tolerability of Betaseron® 500 mcg Subcutaneously Every Other Day and Betaseron® 250 mcg Subcutaneously Every Other Day in Patients With Relapsing-remitting Multiple Sclerosis (RRMS)
Brief Title: Extension of Prior Study Evaluating Safety and Tolerability of Two Doses of Betaseron® to Treat Relapsing-remitting Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 91272; 307320 (Other: Company internal); Beyond (Other: Company internal)
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Results first posted 2009-07-03 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-04

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Relapsing multiple sclerosis; interferon beta 1b; Betaferon; Betaseron
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- ET: IFNB-1b 250 mcg => 250 mcg (Active Comparator): Extension Treatment 250 mcg continued
  Interventions: Drug: Interferon beta 1b (Betaseron, BAY86-5046)
- ET: IFNB-1b 500 mcg => 250 mcg (Experimental): Extension Treatment 500 mcg reduced to 250 mcg
  Interventions: Drug: Interferon beta 1b (Betaseron, BAY86-5046)
- ET: IFNB-1b 500 mcg => 500 mcg (Experimental): Extension Treatment 500 mcg continued
  Interventions: Drug: Interferon beta 1b (Betaseron, BAY86-5046)
- ET: IFNB-1b 250 mcg => 500 mcg (Experimental): Extension Treatment 250 mcg increased to 500 mcg
  Interventions: Drug: Interferon beta 1b (Betaseron, BAY86-5046)

INTERVENTIONS:
Drug: Interferon beta 1b (Betaseron, BAY86-5046) — 250 mcg administered s.c.(subcutaneous) every other day
  Other Names: Betaferon
  Arms: ET: IFNB-1b 250 mcg => 250 mcg
Drug: Interferon beta 1b (Betaseron, BAY86-5046) — 250 mcg administered s.c. every other day (for patients having received 500 mcg before)
  Other Names: Betaferon
  Arms: ET: IFNB-1b 500 mcg => 250 mcg
Drug: Interferon beta 1b (Betaseron, BAY86-5046) — 500 mcg administered s.c. every other day
  Other Names: Betaferon
  Arms: ET: IFNB-1b 500 mcg => 500 mcg
Drug: Interferon beta 1b (Betaseron, BAY86-5046) — 500 mcg administered s.c. every other day (for patients having received 250 mcg before)
  Other Names: Betaferon
  Arms: ET: IFNB-1b 250 mcg => 500 mcg

SUMMARY:
The purpose of this study is to determine if a higher dose of study drug is more effective in preventing relapses in patients with Multiple Sclerosis.

DETAILED DESCRIPTION:
This study has previously been posted by Berlex, Inc. Berlex, Inc. has been renamed to Bayer HealthCare Pharmaceuticals, Inc.

Bayer HealthCare Pharmaceuticals, Inc.is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated statement of informed consent
* Completion of Protocol 307000A
* Negative serum pregnancy test results
* Agreement to adequate contraception, for female patients

Exclusion Criteria:

* Pregnancy or lactation
* History of alcohol or drug abuse
* Inability to administer subcutaneous injections either by self or by caregiver
* Medical, psychiatric or other conditions that compromise the patient's ability to give informed consent, to understand the patient information, to comply with the study protocol, or to complete the study
* Any significant change in the patient's medical condition after enrollment in Study 307000A which would have lead to his/her exclusion from participation that study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2003-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (15):
- United States (15):
  - Los Angeles, California
  - San Francisco, California
  - Washington D.C., District of Columbia
  - Atlanta, Georgia
  - Chicago, Illinois
  - Kansas City, Kansas
  - Louisville, Kentucky
  - Ann Arbor, Michigan
  - Reno, Nevada
  - Stony Brook, New York
  - Durham, North Carolina
  - High Point, North Carolina
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients for this multi-center study included only those who completed in a predecessor study. Patients were enrolled at the end of the preceding study, from 03 Jun 2003 until 06 Jun 2003. Patients who interrupted study medication in accordance with the investigator were eligible, provided it did not result in premature End of Study (EOS).
Pre-assignment Details: For the first 10 weeks of this extension study, patients remained on the IFNB-1b dosage assigned in Study 307000A (Core Treatment). At the Week 10 visit, patients were unblinded by the sponsor and given a choice of drug dosage. They could continue on the original doses, 250 or 500 micrograms, or could change to the other dose (Extension Treatment).
Groups:
- CT: IFNB-1b 250mcg: Core Treatment 250 mcg
- CT: IFNB-1b 500mcg: Core Treatment 500 mcg
Period: Core Treatment Period (CT)
Arm/Group | ET: IFNB-1b 250 mcg => 250 mcg | ET: IFNB-1b 500 mcg => 250 mcg | ET: IFNB-1b 500 mcg => 500 mcg | ET: IFNB-1b 250 mcg => 500 mcg | CT: IFNB-1b 250mcg | CT: IFNB-1b 500mcg
Started | 0 | 0 | 0 | 0 | 36 | 27
Completed | 0 | 0 | 0 | 0 | 36 | 25
Not Completed | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 2
Period: Extension Treatment Period (ET)
Arm/Group | ET: IFNB-1b 250 mcg => 250 mcg | ET: IFNB-1b 500 mcg => 250 mcg | ET: IFNB-1b 500 mcg => 500 mcg | ET: IFNB-1b 250 mcg => 500 mcg | CT: IFNB-1b 250mcg | CT: IFNB-1b 500mcg
Started | 16 | 6 | 19 | 20 | 0 | 0
Completed | 8 | 2 | 14 | 14 | 0 | 0
Not Completed | 8 | 4 | 5 | 6 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 4 | 0 | 0
Not completed — ´Other´ not further itemized | 2 | 3 | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ET: IFNB-1b 250 mcg => 250 mcg | ET: IFNB-1b 500 mcg => 250 mcg | ET: IFNB-1b 500 mcg => 500 mcg | ET: IFNB-1b 250 mcg => 500 mcg | Total
Number analyzed (Participants) | 16 | 6 | 19 | 20 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (9.22) | 32.2 (6.79) | 38.8 (7.57) | 39.3 (7.17) | 38.1 (7.98)
Age, Customized [Number; unit: participants]
  >20-30 years | 3 | 2 | 3 | 1 | 9
  >30-40 years | 7 | 3 | 6 | 10 | 26
  >40-50 years | 4 | 1 | 8 | 8 | 21
  >50 years | 2 | 0 | 2 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 3 | 15 | 12 | 44
  Male | 2 | 3 | 4 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability as Defined by the Number of Subjects With Flu-like Syndrome, Fever, Myalgia, Injection Site Reactions, Injection Site Reactions Pain, Asthenia, Headache, Liver Function Abnormalities, and Bone Marrow Function Abnormalities
Description: Outcome measures are given as the number of patients with common toxicity by the Common Toxicity Criteria (CTC). Toxicity grading is: Grade 1: no study drug action recommended, Grade 2: Dose reduction or interruption of study treatment should be considered (grade 2 Lymphocyte toxicity required no study drug action), Grade 3: Dose reduction or interruption should be considered; interruption is recommended, and Grade 4: Interruption of study drug is recommended (Grade 4 laboratory toxicity was reported as a serious adverse event). Liver and bone marrow abnormalities are measured by lab tests.
Time Frame: At End of Study Visit (week 234)
Population: The statistical analysis was descriptive. For Liver Function Toxicity grading, the total number of patients for 250 micrograms (mcg) - 500 mcg group was 19 instead of 20 for all analyses.
Measure: Number; unit: participants
Arm/Group | ET: IFNB-1b 250 mcg => 250 mcg | ET: IFNB-1b 500 mcg => 250 mcg | ET: IFNB-1b 500 mcg => 500 mcg | ET: IFNB-1b 250 mcg => 500 mcg
Number analyzed (Participants) | 16 | 6 | 19 | 20
participants
  Incidence of flu-like syndrome | 1 | 1 | 4 | 7
  Incidence of fever | 1 | 0 | 1 | 0
  Incidence of myalgia | 0 | 0 | 1 | 0
  Incidence of injection site reactions | 2 | 3 | 4 | 3
  Incidence of injection site reactions pain | 0 | 0 | 1 | 0
  Incidence of asthenia | 4 | 1 | 2 | 3
  Incidence of headache | 2 | 0 | 2 | 3
  Incidence of grade 1 toxicity (ALAT) | 4 | 1 | 8 | 9
  Incidence of grade 2 toxicity (ALAT) | 0 | 0 | 0 | 0
  Incidence of grade 3 toxicity (ALAT) | 0 | 0 | 0 | 0
  Incidence of grade 4 toxicity (ALAT) | 0 | 0 | 0 | 0
  Incidence of grade 1 toxicity (ASAT) | 2 | 1 | 8 | 7
  Incidence of grade 2 toxicity (ASAT) | 1 | 0 | 0 | 0
  Incidence of grade 3 toxicity (ASAT) | 0 | 0 | 0 | 0
  Incidence of grade 4 toxicity (ASAT) | 0 | 0 | 0 | 0
  Incidence of grade 1 toxicity (Bilirubin total) | 10 | 4 | 10 | 14
  Incidence of grade 2 toxicity (Bilirubin total) | 0 | 0 | 1 | 0
  Incidence of grade 3 toxicity (Bilirubin total) | 0 | 0 | 0 | 0
  Incidence of grade 4 toxicity (Bilirubin total) | 0 | 0 | 0 | 0
  Incidence of grade 1 toxicity (Leukocytes) | 3 | 3 | 4 | 6
  Incidence of grade 2 toxicity (Leukocytes) | 1 | 0 | 1 | 2
  Incidence of grade 3 toxicity (Leukocytes) | 0 | 0 | 0 | 0
  Incidence of grade 4 toxicity (Leukocytes) | 0 | 0 | 0 | 0
  Incidence of grade 1 toxicity (Lymphocytes) | 0 | 0 | 1 | 5
  Incidence of grade 2 toxicity (Lymphocytes) | 2 | 0 | 1 | 1
  Incidence of grade 3 toxicity (Lymphocytes) | 0 | 0 | 0 | 1
  Incidence of grade 4 toxicity (Lymphocytes) | 0 | 0 | 0 | 0
  Incidence of grade 1 toxicity (Platelets) | 0 | 0 | 0 | 0
  Incidence of grade 2 toxicity (Platelets) | 0 | 0 | 0 | 0
  Incidence of grade 3 toxicity (Platelets) | 0 | 0 | 0 | 0
  Incidence of grade 4 toxicity (Platelets) | 0 | 0 | 0 | 0
  Incidence of grade 1 toxicity (Hemoglobin) | 0 | 0 | 1 | 1
  Incidence of grade 2 toxicity (Hemoglobin) | 0 | 0 | 0 | 0
  Incidence of grade 3 toxicity (Hemoglobin) | 0 | 0 | 1 | 0
  Incidence of grade 4 toxicity (Hemoglobin) | 0 | 0 | 0 | 0

2. Secondary Outcome: Frequency (Number of Patients Per Group Defined by Cut Off Values and Per Treatment Arm) of Neutralizing Antibody (NAb) Titer to IFNB-1b
Description: Serum samples for analysis of NAbs to interferon (IFN) beta-1b were collected in Study 307000A. In the extension study, NAbs were also monitored for information on persistence or resolution. Serum samples of about 6 mL for NAbs were drawn at Weeks 10, 24, 52, 78, 104 130, 156, 182, 208, 234, 260, 286 or the EOS visit. (NU/ml=neutralizing units/ml).
Time Frame: At End of Study Visit (week 234)
Population: For the NAb analyses data were provided for 40 patients instead of 61 for week 234. Twenty-one patients had no data at this visit.The entries in the table are the number of patients with positive titer in the extension treatment cohorts for the three cutoff titer values. The analyses provide frequencies of positive titers.
Measure: Number; unit: participants
Arm/Group | ET: IFNB-1b 250 mcg => 250 mcg | ET: IFNB-1b 500 mcg => 250 mcg | ET: IFNB-1b 500 mcg => 500 mcg | ET: IFNB-1b 250 mcg => 500 mcg
Number analyzed (Participants) | 8 | 2 | 15 | 15
participants
  NAbs titer, cut-off value 20 NU/ml (minimum) | 2 | 0 | 5 | 3
  NAbs titer, cut-off value 100 NU/ml (minimum) | 1 | 0 | 2 | 2
  NAbs titer, cut-off value 400 NU/ml (minimum) | 1 | 0 | 1 | 1

ADVERSE EVENTS:
Arm/Group | ET: IFNB-1b 250 mcg => 250 mcg | ET: IFNB-1b 500 mcg => 250 mcg | ET: IFNB-1b 500 mcg => 500 mcg | ET: IFNB-1b 250 mcg => 500 mcg
Serious Adverse Events (participants affected / at risk) | 2/16 | 0/6 | 9/19 | 4/20
Other Adverse Events (participants affected / at risk) | 15/16 | 6/6 | 19/19 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ET: IFNB-1b 250 mcg => 250 mcg (N=16) | ET: IFNB-1b 500 mcg => 250 mcg (N=6) | ET: IFNB-1b 500 mcg => 500 mcg (N=19) | ET: IFNB-1b 250 mcg => 500 mcg (N=20)
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 1 | 0
Fever (General disorders) | 0 | 0 | 1 | 0
Necrosis (General disorders) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Surgery (Surgical and medical procedures) | 0 | 0 | 1 | 0
Cerebral Ischemia (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0 | 1 | 0
Myocardial Infarct (Cardiac disorders) | 0 | 0 | 1 | 0
Occlusion (Vascular disorders) | 0 | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Peripheral Vascular Disorder (Vascular disorders) | 0 | 0 | 1 | 0
Pulmonary Embolus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal Disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Joint Disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Grand Mal Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 0
Multiple Sclerosis (Nervous system disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Lung Edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Breast Enlargement (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Otitis Media (Infections and infestations) | 1 | 0 | 0 | 0
Endometrial Disorder (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Kidney Calculus (Renal and urinary disorders) | 1 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ET: IFNB-1b 250 mcg => 250 mcg (N=16) | ET: IFNB-1b 500 mcg => 250 mcg (N=6) | ET: IFNB-1b 500 mcg => 500 mcg (N=19) | ET: IFNB-1b 250 mcg => 500 mcg (N=20)
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 3 | 1
Abscess (Infections and infestations) | 0 | 0 | 1 | 1
Accidental Injury (Injury, poisoning and procedural complications) | 1 | 0 | 4 | 3
Allergic Reaction (Immune system disorders) | 1 | 0 | 3 | 2
Ashthenia (General disorders) | 4 | 1 | 2 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 2
Chills (General disorders) | 0 | 0 | 3 | 0
Cyst (General disorders) | 1 | 0 | 3 | 1
Face Edema (General disorders) | 0 | 0 | 1 | 0
Fever (General disorders) | 1 | 0 | 0 | 0
Flu Syndrom (Infections and infestations) | 1 | 1 | 4 | 7
Heaviness in Extremities (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Hernia (General disorders) | 0 | 0 | 1 | 1
Hormone Level altered (Investigations) | 0 | 0 | 2 | 0
Infection (Infections and infestations) | 2 | 0 | 2 | 3
Laboratory Test abnormal (Investigations) | 0 | 0 | 2 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Pain (General disorders) | 2 | 2 | 4 | 5
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 5 | 3
Pelvic Pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Surgery (Surgical and medical procedures) | 0 | 0 | 1 | 2
Cardiomegaly (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiovascular Disorder (Cardiac disorders) | 0 | 0 | 1 | 0
Cerebral Infarct (Nervous system disorders) | 0 | 0 | 1 | 0
Chest Pain (General disorders) | 1 | 0 | 2 | 0
Hypertension (Vascular disorders) | 2 | 0 | 2 | 3
Migraine (Nervous system disorders) | 1 | 0 | 4 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Peripheral Vascular Disorder (Vascular disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1
Vascular Disorder (Vascular disorders) | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 3 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 1 | 4
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Esophageal Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fecal Incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 3 | 1
Ginigivitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gum Disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Increased Salivation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 4 | 3
Rectal Bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peridontal Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Rectal Disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Tongue Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Tooth Caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Tooth Disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Adrenal Disorder (Endocrine disorders) | 0 | 0 | 1 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Goiter (Endocrine disorders) | 0 | 0 | 1 | 1
Hypothyreodism (Endocrine disorders) | 0 | 0 | 2 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1
Decreased Hemoglobin (Investigations) | 0 | 0 | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 3
Normocytic Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Platelet Count decreased (Investigations) | 0 | 0 | 0 | 1
Injection Site Abscess (Infections and infestations) | 0 | 0 | 1 | 0
Injection Site Necrosis (General disorders) | 0 | 0 | 0 | 1
Injection Site Pain (General disorders) | 0 | 0 | 1 | 0
Injection Site Reaction (General disorders) | 2 | 3 | 4 | 3
Avitaminosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Edema (General disorders) | 0 | 0 | 1 | 0
Gamma-GT increased (Investigations) | 0 | 0 | 1 | 3
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 1
Hyperlipemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Peripheral Edema (General disorders) | 1 | 0 | 2 | 0
SGOT increased (Investigations) | 0 | 0 | 0 | 1
SGPT increased (Investigations) | 0 | 0 | 0 | 2
Uremia (Renal and urinary disorders) | 0 | 0 | 1 | 0
Weight Gain (Investigations) | 2 | 0 | 1 | 1
Weight Loss (Investigations) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bone Disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Bone Fracture (not spontaneous) (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint Disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myasthenia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3 | 7
Tendon Disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Abnormal Gait (General disorders) | 0 | 0 | 0 | 2
Amnesia (Nervous system disorders) | 1 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 2 | 1 | 2 | 2
Ataxia (Nervous system disorders) | 4 | 0 | 1 | 2
Confusion (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 4 | 3 | 4 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 3 | 2
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0
Emotional Lability (Psychiatric disorders) | 0 | 1 | 0 | 0
Foot Drop (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 2 | 3
Hot Flashes (Vascular disorders) | 1 | 0 | 0 | 0
Hypalgesia (Nervous system disorders) | 1 | 0 | 3 | 0
Hyperkinesia (Nervous system disorders) | 1 | 0 | 0 | 0
Hypertonia (Nervous system disorders) | 3 | 0 | 3 | 1
Hypesthesia (Nervous system disorders) | 5 | 3 | 7 | 9
Incoordination (Nervous system disorders) | 2 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 3 | 4
Libido decreased (Psychiatric disorders) | 0 | 0 | 1 | 0
Multiple Sclerosis (Nervous system disorders) | 4 | 3 | 2 | 6
Nervousness (Psychiatric disorders) | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 2 | 2
Neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 2 | 0 | 1 | 3
Ophthalmoplegia (Eye disorders) | 0 | 0 | 0 | 1
Paresthesia (Nervous system disorders) | 5 | 3 | 7 | 5
Reflexes decreased (Nervous system disorders) | 0 | 0 | 1 | 1
Reflexes increased (Nervous system disorders) | 1 | 0 | 1 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 1 | 0
Speech Disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Sweating increased (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Thinking abnormal (Psychiatric disorders) | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 1 | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0 | 2
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 4 | 1 | 3 | 2
Cough increased (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal Septum Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 1
Pleural Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 3
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 2 | 1 | 5 | 5
Upper Respiratory Infection (Infections and infestations) | 5 | 1 | 2 | 7
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Breast Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Female Lactation (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Fungal Dermatitis (Infections and infestations) | 0 | 0 | 2 | 0
Petechial Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Skin Benign Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Skin Discoloration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin Disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3
Skin Necrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Blurred Vision (Eye disorders) | 2 | 0 | 2 | 5
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 1 | 0
Ear Disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Ear Pain (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Eye Disorder (Eye disorders) | 0 | 1 | 0 | 0
Eye Pain (Eye disorders) | 0 | 0 | 3 | 1
Optic Neuritis (Nervous system disorders) | 0 | 0 | 1 | 0
Otitis Media (Infections and infestations) | 1 | 0 | 1 | 0
Ptosis (Eye disorders) | 0 | 0 | 1 | 0
Pupillary Disorder (Eye disorders) | 0 | 0 | 0 | 1
Refraction Disorder (Eye disorders) | 1 | 0 | 0 | 0
Retinal Disorder (Eye disorders) | 1 | 0 | 0 | 0
Taste Perversion (Nervous system disorders) | 0 | 0 | 1 | 0
Visual Field Defect (Nervous system disorders) | 1 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Dyspareunia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Genital Leukoplakia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Impotence (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Increased Urinary Frequency (Renal and urinary disorders) | 1 | 1 | 0 | 0
Kidney Calculus (Renal and urinary disorders) | 0 | 0 | 2 | 0
Leukorrhea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Menstrual Disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Papanicolaou Smear suspicious (Investigations) | 0 | 0 | 0 | 1
Urethritis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 2
Urinary Retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary Tract Disorder (Renal and urinary disorders) | 0 | 0 | 1 | 1
Urinary Tract Infection (Infections and infestations) | 4 | 0 | 6 | 3
Urinary Urgency (Renal and urinary disorders) | 1 | 1 | 0 | 1
Urination impaired (Renal and urinary disorders) | 0 | 1 | 1 | 1
Vaginitis (Infections and infestations) | 0 | 0 | 1 | 0
Vulvovaginal Disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The 40 patients in the NAb frequency summaries are the total number of patients with NAb titers at week 234. Official HARTS-to-MedDRA Mapping was used.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No